CLINICAL TRIAL: NCT05506644
Title: A Proof-of-Concept Study Exploring HRV-Biofeedback for Psoriasis and Associated Psychological Comorbidities
Brief Title: Biofeedback for Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bastyr University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1714
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Psoriasis; Psoriasis Vulgaris; Psychophysiological Disorder; Anxiety; Depression; Psychological Stress; Physiological Stress; Quality of Life; Skin Disorder; Skin Diseases
Keywords: Psoriasis; Anxiety; Depression; Biofeedback; Stress; Psychophysiological Disorder; Skin Disease
MeSH Terms: conditions — Psoriasis; Psychophysiologic Disorders; Anxiety Disorders; Depression; Stress, Psychological; Skin Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRV-Biofeedback (Experimental)
  Interventions: Other: HRV-Biofeedback/Mind-Body Therapy

INTERVENTIONS:
Other: HRV-Biofeedback/Mind-Body Therapy — A 7-week protocol using real-time feedback on heart rate variability

SUMMARY:
We are conducting a proof-of-concept trial to study the impact of HRV-biofeedback, a mind-body technique designed to improve stress resilience, on the quality of life, mood, and clinical skin severity of patients with psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a common, chronic stress-related disease of the skin and joints that is associated with significantly impaired quality of life (QoL) and psychological comorbidity, most notably anxiety, depression, and suicidality. The objective of this study is to explore the influence of heart rate variability-biofeedback training (HRV-BF) on measures rating QoL, mental health, and clinical severity of psoriasis. We aim to further understand the bidirectional relationship between stress and the skin and to determine whether HRV-BF has the potential to be a beneficial adjuvant therapy for psychocutaneous disorders. A single-arm, proof-of-concept trial will be conducted using a modified, 7-week HRV-BF resiliency protocol at Bastyr University California in a small sample of subjects with moderate to severe plaque psoriasis. In order to measure the outcomes of the intervention on the clinical manifestations of psoriasis, we will be administering a set of validated, physician-rated and patient-reported questionnaires, including the Psoriasis Area and Severity Index (PASI), Dermatology Life Quality Index (DLQI), Patient Health Questionnaire (PHQ-9), and Generalized Anxiety Disorder (GAD-7), in addition to other HRV-BF-specific screening questionnaires to assess whether the subject has any contraindications to this protocol. These assessments will be collected at baseline, end of trial, and at 1-month follow-up for statistical analysis. The goal of this trial is to explore the novel application of HRV-BF for psychocutaneous disorders in order to fill a gap in the provision of evidence-based, integrative services addressing the serious and sometimes fatal psychological impacts of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosed with or are currently experiencing symptoms of psoriasis
* Located in San Diego or within driving distance
* Have daily access to a smart phone, computer, or tablet
* Able to read and understand English

Exclusion Criteria:

* High risk of suicidality
* History of chronic kidney disease
* Pacemaker
* Active pregnancy or treatment of cancer or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Life Quality Index | 11 weeks
Dermatology Life Quality Index | 11 weeks
Generalized Anxiety Disorder-7 | 11 weeks
Patient Health Questionnaire-9 | 11 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bastyr University Clinic, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No